CLINICAL TRIAL: NCT03262441
Title: Mycophenolate Mofetil Therapy for Reduction of the HIV Reservoir
Brief Title: MMF for HIV Reservoir Reduction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Joshua Schiffer, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8589; STUDY00002182 (Other: University of Washington IRB); 109614-62-RGRL (Other Grant/Funding Number: American Foundation for AIDS Research); ACTU-2100 (Other: University of Washington)
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Human Immunodeficiency Virus I Infection
Keywords: HIV; Antiretroviral treatment; Mycophenolate mofetil; Cure; Latency; Reservoir; CD4 T cell; Anti-proliferation
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized pilot trial to determine whether MMF given over 22 months meaningfully decreases the size of the HIV reservoir. Study participants will be followed closely for at least 22 months with safety labs and serial measurements of the HIV reservoir (specifically, cell-associated HIV DNA and mRNA (ca-DNA & ca-RNA), quantitative viral outgrowth assay (QVOA), and single copy plasma viral load (scVL)). "Go/no-go" decision will occur after 12 months based on pre-defined thresholds of reduction in the HIV reservoir measured with ca-DNA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mycophenolate mofetil (Experimental): Mycophenolate Mofetil 500mg Tablets once per day for one week as a lead in to limit drug-related side effects. Provided they are tolerating the drug at lower dose, they will then initiate Mycophenolate Mofetil 500mg Tablets twice daily orally for 22 months
  Interventions: Drug: Mycophenolate Mofetil 500Mg Tab

INTERVENTIONS:
Drug: Mycophenolate Mofetil 500Mg Tab — 500 mg once daily for one week. If tolerating the drug, then initiate twice daily for 22 months
  Other Names: Mycophenolate Mofetil Tablets USP Roxane Laboratories

SUMMARY:
This is an open label, randomized Phase II study to determine whether Mycophenolate mofetil (MMF) given over 22 months meaningfully decreases the size of participants' HIV reservoir.

In addition to primary safety endpoints, the following hypotheses regarding drug efficacy will be tested:

1. MMF will be well tolerated and will not decrease adherence to or antiviral efficacy of ART.
2. Peripheral CD4+ T-cell counts and percentages will not meaningfully decrease during treatment with MMF and ART.
3. There will be no excess risk of opportunistic infections in MMF-treated study participants.
4. MMF therapy will lead to a progressive decrease in reservoir size over 22 months of treatment.
5. MMF therapy will lead to a continual shift in HIV reservoir composition from primarily effector memory CD4+ T cells (TEM) and central memory CD4+ T cells (TCM), to primarily stem cell like memory (TSCM) and naïve (TN) CD4+ T cells.
6. MMF will eliminate detectable measures of the HIV reservoir, including by cell-associated DNA/mRNA and quantitative viral outgrowth.
7. MMF will not decrease the humoral immune response to routine annual influenza vaccination.

DETAILED DESCRIPTION:
This is an open-label, randomized pilot trial to determine whether MMF given over 22 months meaningfully decreases the size of the HIV reservoir.

At the University of Washington in Seattle, investigators will enroll 5 study participants who have been on ≥2 years of suppressive ART. Study participants will be followed closely for at least 22 months with safety labs and serial measurements of the HIV reservoir (specifically, cell-associated HIV DNA and mRNA (ca-DNA & ca-RNA), quantitative viral outgrowth assay (QVOA), and single copy plasma viral load (scVL)). A "go/no-go" decision will occur after 12 months based on pre-defined thresholds of reduction in the HIV reservoir measured with ca-DNA.

All participants will be offered enrollment in a sub-study in which an anoscopy with rectum biopsies is performed on 3 occasions to assess the reservoir in the gastrointestinal lymphatic tissue (GALT).

Investigators will vaccinate study participants with the annual influenza vaccine and analyze their humoral response to this vaccine approximately one month later with a routine blood draw done in conjunction with a safety labs blood draw.

Investigators hypothesize that low doses of MMF will be well tolerated among healthy HIV-infected study participants who have fully ART-suppressed HIV. Investigators hypothesize that the incidence of opportunistic infections will not exceed that of comparable larger cohorts of HIV-treated patients. Of note, certain opportunistic infections such as herpes zoster or HSV-2 recurrence continue to occur despite suppressive ART, while pneumocystis pneumonia, CMV end organ disease, cryptococcus and many other opportunistic infections are much less common in this context. Therefore, in the event of an infection, Investigators will confer with the data safety management (DSM) panel to discuss whether this event is directly attributable to MMF. Finally, investigators hypothesize that peripheral blood CD4+ and CD8+ T cell counts will remain unchanged throughout MMF therapy, and that HIV replication will remain controlled on ART with addition of MMF.

Investigators hypothesize at least a 0.25-log reduction in cell-associated HIV DNA at one-year intervals in study participants who have a demonstrated anti-proliferative response to MMF treatment. Investigators hypothesize that cell-associated HIV DNA will undergo a shift from predominant residence in TCM and TEM to predominant residence in TN and TSCM. In regards to our sub-study, investigators predict that reservoir depletion will occur with equivalent rates in blood and GALT.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV infection, by two different positive antibody tests and/or detectable plasma HIV RNA on two different dates
2. ≥18 and ≤65 years of age
3. Continuous ART during the last two years, with current ART preferably including an integrase inhibitor
4. HIV RNA <40 copies / mL on four occasions during continuous ART of ≥ 2 years with no more than one blip of <1000 HIV RNA copies / mL
5. CD4+ T cell count > 350/mm3 within the past 365 days
6. Karnofsky score ≥80
7. Plan to reside in area 2 years
8. Consents to study
9. Tolerability of MMF during one week dose escalation lead-in phase of 500 mg once daily
10. Demonstrated anti-proliferative effect of MMF 500 mg twice daily

Exclusion Criteria:

1. Active malignancy including skin cancer, myelodysplastic syndrome, or myeloproliferative disease within 24 weeks prior to study entry
2. Prior organ or bone marrow transplantation
3. Diagnosed autoimmune disease
4. Medical need for ongoing treatment with an immunosuppressive drug
5. Diagnosis of AIDS (defined as any AIDS-defining opportunistic infection or cancer, or a history of blood CD4+ T cell count < 200/µL)
6. Active opportunistic infection
7. Using disallowed medications (see 4.3)
8. Vomiting or diarrhea which prohibits consistent use of study drugs
9. Pregnant, intention to become pregnant, or breastfeeding
10. Woman of child bearing age who are NOT using two forms of birth control OR practicing complete abstinence
11. Excessive ingestion of ethanol, determined by an AUDIT score of >8
12. Substance abuse
13. History of medical non-compliance
14. Quantiferon TB positive
15. The following laboratory values (< 30 days before enrollment):

    * Hemoglobin < 8.5 mg/dL
    * Absolute neutrophil count < 1000 cells/mm3
    * ALT > 2 x upper limit of normal
    * Platelet count < 100,000/uL
    * Creatinine clearance < 60 mL/min

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua T Schiffer, MD MSc, Principal Investigator — Fred Hutchinson Cancer Center; Florian Hladik, MD PhD, Principal Investigator — University of Washington
Locations (1):
- 2 West Clinic at Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reeves DB, Duke ER, Hughes SM, Prlic M, Hladik F, Schiffer JT. Anti-proliferative therapy for HIV cure: a compound interest approach. Sci Rep. 2017 Jun 21;7(1):4011. doi: 10.1038/s41598-017-04160-3. PMID 28638104
- [Derived] Schiffer JT, Levy C, Hughes SM, Pandey U, Padullo M, Jerome KR, Zhu H, Puckett K, Helgeson E, Harrington RD, Hladik F. Stable HIV Reservoir Despite Prolonged Low-Dose Mycophenolate to Limit CD4+ T-cell Proliferation. Open Forum Infect Dis. 2022 Nov 19;9(12):ofac620. doi: 10.1093/ofid/ofac620. eCollection 2022 Dec. PMID 36519118

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the University of Washington AIDS Clinical Trials Unit at Harborview Medical Center in Seattle. The first participant enrolled February 12, 2018 and the last participant enrolled in August 14, 2018.
Period: Overall Study
Arm/Group | Mycophenolate Mofetil
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mycophenolate Mofetil
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Cell-associated HIV DNA (Ca-DNA) Levels Per 10^6 T Cells Over 12 Months
Description: Regression slope of change in cell-associated HIV DNA (ca-DNA) as measured by multiplexed digital droplet PCR in study participants on MMF calculated from 4 time points between 0 & 12 months
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: log10 caDNA copies per 10^6 T-cells/week
Arm/Group | Mycophenolate Mofetil
Number analyzed (Participants) | 4
log10 caDNA copies per 10^6 T-cells/week | -0.00033 [-0.0020 to 0.0014]
Statistical Analysis 1: Comparison: Mycophenolate Mofetil; Test type: Other; Slope = -0.00033, 95% CI 2-sided [-0.0020 to 0.0014]

2. Primary Outcome: Change in Cell-associated HIV DNA (Ca-DNA) Levels Per 10^6 Effector Memory CD4+ T Cells Over 12 Months
Description: Regression slope of change in cell-associated HIV DNA (ca-DNA) as measured by multiplexed digital droplet PCR in study participants on MMF calculated from 3 time points between 0 & 12 months
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: log10 caDNA copies per 10^6 T-cells/week
Arm/Group | Mycophenolate Mofetil
Number analyzed (Participants) | 4
log10 caDNA copies per 10^6 T-cells/week | 0.001 [-0.0036 to 0.0056]
Statistical Analysis 1: Comparison: Mycophenolate Mofetil; Test type: Other; Slope = 0.001, 95% CI 2-sided [-0.0036 to 0.0056]

3. Primary Outcome: Change in Cell-associated Intact HIV DNA (Ca-iDNA) Levels Per 10^6 T Cells Over 12 Months
Description: Regression slope of change in cell-associated intact HIV DNA (ca-iDNA) as measured by multiplexed digital droplet PCR in study participants on MMF calculated from 4 time points between 0 & 12 months
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: log10 caDNA copies per 10^6 T-cells/week
Arm/Group | Mycophenolate Mofetil
Number analyzed (Participants) | 4
log10 caDNA copies per 10^6 T-cells/week | .0024 [-0.0030 to 0.0078]
Statistical Analysis 1: Comparison: Mycophenolate Mofetil; Test type: Other; Slope = 0.0024, 95% CI 2-sided [-0.003 to 0.0078]

4. Secondary Outcome: Blood CD4+ T Cells Per mm^3 Blood
Description: Frequency of participants with any time point with <200 CD4+ T cells per mm^3 from 4 sampled time points between 0 & 12 months
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil
Number analyzed (Participants) | 4
participants | 0

5. Secondary Outcome: Incidence of Opportunistic Infection
Description: Number of participants experiencing opportunistic infection
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil
Number analyzed (Participants) | 4
participants | 0

ADVERSE EVENTS:
Time Frame: 20 months
Arm/Group | Mycophenolate Mofetil
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mycophenolate Mofetil (N=5)
Finger cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a small and uncontrolled study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT03262441/Prot_SAP_000.pdf